CLINICAL TRIAL: NCT07369674
Title: Epidemiological and Clinical Characteristics of Patients With Hepatic Hydatid Cysts in an Endemic Area: A Multi-Center Investigation in Najaf City, Iraq.
Brief Title: Epidemiological Study of Hydatid Cyst in Najaf City, Iraq
Acronym: Hydatid cyst
Status: Completed | Type: Observational
Sponsor: Al-Kafeel University (Other)
Responsible Party: Principal Investigator, Samer Al Hakkak, Dean, Al-Kafeel University
Other Study IDs: University of Alkafeel; self (Other: University of Alkafeel)
Record Dates: First submitted 2026-01-05; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hydatid Cyst, Hepatic
MeSH Terms: conditions — Echinococcosis, Hepatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 350 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Cystic echinococcosis (hydatid cyst) is a significant zoonotic disease endemic to Iraq. Understanding the localized clinical and epidemiological trends is vital for improving surgical outcomes and public health strategies.

Objective To determine the epidemiological and clinical profile of patients diagnosed with liver hydatid cysts within the hospitals of Najaf City, Iraq.

DETAILED DESCRIPTION:
Patients and Methods This retrospective observational study analyzed the records of 350 patients treated for liver hydatid cysts across multiple hospitals in Najaf, Iraq, from February 2021 to June 2024. Data were extracted from official patient records, including sociodemographic characteristics, clinical presentation, cyst morphology, and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

All patients of any age or gender with a radiologically or surgically confirmed diagnosis of liver hydatid cyst

Exclusion Criteria:

Patients with hydatid cysts located exclusively in extra-hepatic sites (e.g., brain, lung, bone, spleen, or muscle). Patients with severe chronic comorbidities or incomplete medical records were also excluded to ensure data integrity

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective, observational study was conducted on a total of 350 patients diagnosed with liver hydatid cysts. The study was carried out at multiple centers in Najaf City, Iraq, including major governmental surgical hospitals and specialized centers, covering the period from February 2021 to June 2024.
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
To determine the epidemiological and clinical profile of patients diagnosed with liver hydatid cysts within the hospitals of Najaf City, Iraq. | February 2021 to June 2024
  This retrospective observational study analyzed the records of 350 patients treated for liver hydatid cysts across multiple hospitals in Najaf, Iraq, from February 2021 to June 2024.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alkafeel, Najaf, Iraq

IPD SHARING:
Plan to Share IPD: Undecided
undecided